CLINICAL TRIAL: NCT01307644
Title: Web-Based Weight Loss & Weight Maintenance Intervention for Older Rural Women
Brief Title: Web-Based Weight Loss & Weight Maintenance Intervention for Older Rural Women, Also Known as Women Weigh-in for Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0237-10-FB; 1R01NR010589-01A2 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Rural Health; Weight Loss; Weight Maintenance; Rural Middle Aged and Older Women; Web Intervention Weight Loss; Class I, II, & III obese (BMI 28 to 45)
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Web-based only (WO) weight intervention (Experimental): A comprehensive lifestyle modification intervention for healthy eating and activity delivered by web only to facilitate Phase I weight loss (weekly messages baseline to 6 months), Phase 2 guided weight loss and weight maintenance (bi-weekly hot topics news, 6-18 months) and Phase 3 self-managed weight maintenance (6 monthly and 3 bi-monthly new content, 18-30 months).
  Interventions: Behavioral: Experimental: Web-based only (WO) weight intervention
- WO & peer-led discussion board (WD) (Experimental): Includes WO intervention, including all 3 Phases for weight loss and weight maintenance, supplemented with peer-lead discussion board. A peer leader will facilitate the asynchronous discussion group. The primary purpose of this group is to provide support, increase self-efficacy (role modeling by successful women and leader) and discuss progress toward goals.
  Interventions: Behavioral: Experimental: Web-based only (WO) weight intervention; Behavioral: Experimental: WO plus peer-led discussion board (WD)
- WO & professional email counseling (WE) (Experimental): Includes WO intervention, including all 3 Phases for weight loss and weight maintenance, supplemented with professional email-counseling by experienced counselor who will review women's web-logs of eating, activity, weight and goal-setting on web-site and send e-mail feedback.
  Interventions: Behavioral: Experimental: Web-based only (WO) weight intervention; Behavioral: Experimental: WO & professional email counseling (WE)

INTERVENTIONS:
Behavioral: Experimental: Web-based only (WO) weight intervention — The WO intervention included evidence-based lifestyle modification for healthy eating and activity, with self-monitoring and goal setting, and messages based on constructs from the Health Promotion Model across 3 phases. The intent of the phases was to deliver more intensive intervention during Phase 1, transitioning to less intensive intervention during phase 2, to providing support for self managed weight maintenance during Phase 3.
Behavioral: Experimental: WO plus peer-led discussion board (WD) — Includes WO intervention plus asynchronous discussion board managed by peer leader, whose identity is masked. The peer leader who posted theme-based messages, called primers, that were consistent with WO themes across phases.
  Arms: WO & peer-led discussion board (WD)
Behavioral: Experimental: WO & professional email counseling (WE) — Includes WO intervention plus professional email counseling provided by a registered dietitian whose identity is masked. The email counselor is responsible for reviewing eating, activity, weight logs, and goals on the web-site and send e-mail feedback, in addition to responding to email questions. The e-mail process will follow the 5A's Model for Behavioral Counseling (assess, advise, agree, assist, and arrange) that was adapted for this study.
  Arms: WO & professional email counseling (WE)

SUMMARY:
This project will evaluate an Internet delivery strategy to address weight loss and maintenance among rural midlife and older women.

DETAILED DESCRIPTION:
According to the National Institutes of Health, "obesity is one of the most daunting health challenges of the 21st century". Approximately 2/3 of all adults are overweight or obese. Efforts to abate the growing prevalence of obesity have not been successful. The Strategic Plan for NIH Obesity Research proposes preventing and treating obesity through lifestyle modification. The purpose of this study is to evaluate the effectiveness of a theory-based intervention framed within the Health Promotion Model (HPM) in facilitating weight loss and maintenance through promotion of healthy eating and physical activity among an underserved, vulnerable population of overweight or obese rural women aged 40-69. During these years, women experience increases in peri- and post-menopausal health risks that are magnified if they are overweight or obese. Weight loss will reduce risks and enhance functional status as they age. Maintenance of weight loss will be emphasized. The Internet offers a way to reach isolated rural women who have limited options for weight loss guidance. PUBLIC HEALTH RELEVANCE: Obesity is recognized as a major and growing public health problem. While many weight loss programs have been successful in the short term, they have not been successful in helping to maintain weight loss.

ELIGIBILITY:
Inclusion Criteria:

* women aged 40-69
* overweight or Class I & II obese (BMI 28 to 39.9)or BMI 40 to 45 with physician clearance
* state a commitment to losing weight
* speak and read English
* able to communicate over the telephone
* able to use a computer with minimal assistance and complete electronic forms and surveys
* have access to and are able to access the Internet
* commitment to access the website as required by the research intervention including weekly self-reporting of calories and fat grams, weekly self-reporting of physical activity, pedometer steps, and body weight, and weekly (or more often) participation in other website components as determined by group to which randomized and phase of intervention
* have or are willing to obtain an email account
* have access to a DVD player
* able to walk without an assistive device
* answer 'no' to all questions on the Physical Activity Readiness Questionnaire (PAR-Q) or obtain clearance from their physician to become more active

Exclusion Criteria:

* diagnosed with Type 1 diabetes
* diagnosed with Type 2 diabetes and require insulin
* ≥ 10% weight loss in last six months
* enrolled in a weight loss management program
* enrolled in a formal program of cardiac rehabilitation or undergoing physical rehabilitation
* taking medications that affect weight loss or weight gain
* other physical or medical restrictions that would preclude following the minimum recommendations for moderate physical activity and healthy eating.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
1: Differences in Change in Weight between Groups - Body Weight (kg) | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 1: The primary aim of the study was to compare the effectiveness of web-based only (WO) intervention with web-based interventions supplemented with peer-led discussion support group (WD) or professional email counseling (WE) for achieving change in the primary outcome of body weight between groups across three phases [Phase I guided weight loss (baseline to 6 months), Phase 2 continued guided weight loss and weight maintenance over 12 months (6 months and 18 months), Phase 3 self-directed weight maintenance over 12 months (18 months and 30 months)].
Differences in Change in Weight between Groups - waist circumference (cm) | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 1: Differences in Change in Weight between Groups - waist circumference (cm)
Differences in Change in Healthy Eating and Activity Outcomes between Groups - Kcal intake | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: The secondary aim of the study was to compare the effectiveness of web-based only (WO) intervention with web-based interventions supplemented with peer-led discussion support group (WD) or professional email counseling (WE) for achieving change in primary outcomes of behavioral and biomarkers of healthy eating and activity between groups across three phases [Phase I guided weight loss (baseline and 6 months), Phase 2 continued guided weight loss and weight maintenance over 12 months (6 months and 18 months), Phase 3 self-directed weight maintenance over 12 months (18 months and 30 months)]
Differences in Change in Healthy Eating and Activity Outcomes between Groups - Weekly minutes moderate or greater intensity activity | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: Differences in Change in Healthy Eating and Activity Outcomes between Groups - Weekly minutes moderate or greater intensity activity
Differences in Change in Healthy Eating and Activity Outcomes between Groups - Blood Pressure | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: Differences in Change in Healthy Eating and Activity Outcomes between Groups - Blood Pressure
Differences in Change in Healthy Eating and Activity Outcomes between Groups - Blood Lipids | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: Differences in Change in Healthy Eating and Activity Outcomes between Groups - Blood Lipids

SECONDARY OUTCOMES:
Differences in Change in attaining Criterion-based Weight loss targets between Groups | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 1: Differences in Change in attaining Criterion-based Weight loss targets between Groups
Differences in Change in attaining Criterion-based Healthy Eating between Groups | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: Differences in Change in attaining Criterion-based Healthy Eating between Groups
Differences in Change in attaining Criterion-based Physical Activity between Groups | Phase 1-baseline and 6 months, Phase 2-6 months and 18 months, Phase 3-18 months and 30 months
  Aim 2: Differences in Change in attaining Criterion-based Physical Activity between Groups

CONTACTS AND LOCATIONS:
Overall Officials: Carol H Pullen, EdD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hageman PA, Mroz JE, Yoerger MA, Pullen CH. Weight loss is associated with improved quality of life among rural women completers of a web-based lifestyle intervention. PLoS One. 2019 Nov 19;14(11):e0225446. doi: 10.1371/journal.pone.0225446. eCollection 2019. PMID 31743365
- [Derived] Hageman PA, Mroz JE, Yoerger MA, Pullen CH. User Engagement Associated with Web-Intervention Features to Attain Clinically Meaningful Weight Loss and Weight Maintenance in Rural Women. J Obes. 2019 Mar 3;2019:7932750. doi: 10.1155/2019/7932750. eCollection 2019. PMID 30944736
- [Derived] Hageman PA, Pullen CH, Yoerger M. Physical Function and Health-Related Quality of Life in Overweight and Obese Rural Women Who Meet Physical Activity Recommendations. J Aging Phys Act. 2018 Jul 1;26(3):438-444. doi: 10.1123/japa.2017-0117. Epub 2018 Jun 13. PMID 28952857
- [Derived] Hageman PA, Pullen CH, Hertzog M, Pozehl B, Eisenhauer C, Boeckner LS. Web-Based Interventions Alone or Supplemented with Peer-Led Support or Professional Email Counseling for Weight Loss and Weight Maintenance in Women from Rural Communities: Results of a Clinical Trial. J Obes. 2017;2017:1602627. doi: 10.1155/2017/1602627. Epub 2017 Apr 5. PMID 28480078
- [Derived] Shade MY, Berger AM, Dizona PJ, Pozehl BJ, Pullen CH. Sleep and health-related factors in overweight and obese rural women in a randomized controlled trial. J Behav Med. 2016 Jun;39(3):386-97. doi: 10.1007/s10865-015-9701-y. Epub 2015 Dec 11. PMID 26661065
- [Derived] Hageman PA, Pullen CH, Hertzog M, Boeckner LS, Walker SN. Web-based interventions for weight loss and weight maintenance among rural midlife and older women: protocol for a randomized controlled trial. BMC Public Health. 2011 Jun 30;11:521. doi: 10.1186/1471-2458-11-521. PMID 21718512